CLINICAL TRIAL: NCT03961815
Title: An Open-label, Long-term Extension Study of Brazikumab in Participants With Moderately to Severely Active Crohn's Disease (INTREPID OLE)
Brief Title: Open-label Extension Study of Brazikumab in Crohn's Disease
Acronym: INTREPID OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic decision to discontinue the development of brazikumab in inflammatory bowel disease.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D5271C00002; #3150-303-008 (Other: Legacy); 2019-001866-14 (EudraCT Number)
Record Dates: First submitted 2019-05-08; First posted 2019-05-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Crohn's Disease; IBD
Keywords: Crohn's Disease; Inflammatory bowel disease; Brazikumab; IL23 receptor; IBD; CD
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brazikumab Induction Dose (Experimental): Administer at Week 0, Week 4, and Week 8
  Interventions: Drug: Brazikumab Induction Dose
- Brazikumab Maintenance Dose (Experimental): Administer at 4-week intervals through Week 52 Participants who receive IV induction dosing will be administered brazikumab SC at 4-week intervals starting Week 12 through Week 52
  Interventions: Drug: Brazikumab Maintenance Dose

INTERVENTIONS:
Drug: Brazikumab Induction Dose — Participants who met criteria for early termination due to lack of efficacy (rescue treatment criteria) or who did not meet CDAI response at Week 52 in the lead-in study D5121C00001 are considered inadequate/non responders, and will receive IV induction dosing brazikumab at Week 0, Week 4, and Week 8 followed by maintenance dosing of brazikumab subcutaneously every 4 weeks thereafter up to Week 52.
  Arms: Brazikumab Induction Dose
Drug: Brazikumab Maintenance Dose — Responders from Lead-In study D5271C00001 who completed requirements through Week 52 and met CDAI response (CDAI score of < 150 points or CDAI reduction from Baseline of ≥ 100 points) without ongoing rescue treatment at Week 52 in the lead-in study. will receive maintenance dose of brazikumab administered subcutaneously every 4 weeks through Week 52, starting at Week 0. The subcutaneous dose of brazikumab will be administered to all responders/completers in the lead-in study regardless of the prior treatment administered
  Arms: Brazikumab Maintenance Dose

SUMMARY:
The purpose of Study D5271C00002 (Legacy #3150-303-008) is to permit participants in D5271C00001 (Legacy #3150-301-008) to receive open-label brazikumab in Study D5271C00002 (Legacy #3150-303-008). This will permit long-term observation of safety in these participants with brazikumab.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants with successful completion or early termination due to lack of efficacy from Study D5271C00001 (Legacy #3150-301-008).

   Meets 1 of the following criteria for successful completion or early termination due to lack of efficacy from Study D5271C00001 (Legacy #3150-301-008):
   1. A participant is considered to have completed the D5271C00001 (Legacy #3150-301-008) study if they have received scheduled study interventions, completed scheduled visits, and completed Week 52 assessments.
   2. A participant in Study D5271C00001 (Legacy #3150-301-008) who discontinued from the study due to lack of efficacy after a minimum of 12 weeks of double-blind treatment and met criteria for the use of rescue treatment in the lead-in protocol.
2. Criterion deleted as part of Amendment.
3. Each participant must have had the ileocolonoscopic procedure at the final visit (Week 52, Week 12, or early termination after Week 12 of Study D5271C00001 (Legacy # 3150-301-008).
4. Female participants of childbearing potential must have a negative urine pregnancy test prior to administration of study intervention and must agree to use a highly effective method of birth control (confirmed by the investigator) from signing the ICF throughout the study duration and for at least 18 weeks after last dose of study intervention.
5. Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if they have been amenorrhoeic for 12 months prior to signing the ICF without an alternative medical cause.
6. Nonsterilized males who are sexually active with a female partner of childbearing potential must comply with the methods of contraception during treatment and until the end of relevant systemic exposure in the male participant, plus a further 18 weeks.
7. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.
8. Written informed consent from the participant has been obtained prior to any study related procedures.
9. Legally authorized representative consent has been obtained (if applicable).
10. Written documentation has been obtained in accordance with the relevant country and local privacy requirements, where applicable.
11. Demonstration of adequate compliance with the study procedures in Study D5271C00001 (Legacy #3150 301-008) in the opinion of the investigator and/or sponsor.
12. Willingness and ability to attend all study visits, comply with the study procedures, read and write in order to complete questionnaires, and be able to complete the study.

Complete inclusion criteria are in the study protocol

Exclusion Criteria:

1. Any participant with an unresolved AE from the Study D5271C00001 (Legacy #3150 301-008) that would limit the participant's ability to participate in or complete this study.
2. Current diagnosis of ischemic colitis, colonic mucosal dysplasia, or primary sclerosing cholangitis.
3. Organ or cell-based transplantation (eg, islet cell transplantation or autologous stem cell transplantation) with the exception of corneal transplant.
4. Any other condition or finding that, in the investigator's or sponsor's opinion, would either confound proper interpretation of the study or expose a participant to unacceptable risk.
5. History of cancer except for basal cell and/or squamous cell carcinoma of the skin, and carcinoma in situ of the cervix within 12 months of screening.
6. Participant meets criteria for discontinuation of study intervention during prior the D5271C00001 (Legacy #3150 301-008) study (excluding lack of efficacy).
7. Criterion deleted as part of Amendment.
8. Known history of primary immunodeficiency, splenectomy, or any underlying condition that predisposes the subject to infection, including HIV infection.
9. Prolonged QTcF interval (QTc >450 msec or QTC >480 for participants with bundle branch block; determined by central ECG), or conditions leading to additional risk for QT prolongation (eg, congenital long-QT syndrome).
10. Clinically significant kidney disease including but not limited to:

    (a) Chronic kidney disease with an estimated glomerular filtration rate of less than 30 ml/min calculated by MDRD equation, as applicable, by the central laboratory at screening are excluded.
11. Participant requires additional immunosuppressive therapy (aside from permitted concomitant medication), biological treatment, or prohibited treatment.
12. Participant received a Bacille Calmette-Guérin vaccination within 12 months of Week 0 (Visit 1) or any other live vaccine < 4 weeks prior to Week 0 (Visit 1) or is planning to receive any such vaccine over the course of the study.
13. Participant received a prohibited medication during participation in the lead-in study or during screening for this study.
14. Participant is planning to receive an investigational drug (other than study intervention) or investigational device at any time during Study D5271C00002 (Legacy #3150-303-008) with the exception of "registry" or "cohort" trials.
15. Participants with a known hypersensitivity to brazikumab or any of the excipients of the product.
16. Protocol-defined abnormal laboratory results at screening. 17. Females who are pregnant, nursing, or planning a pregnancy during the study OR females who are of childbearing potential and do not agree to use a highly effective method of contraception consistently and correctly.

18 Participant is directly or indirectly involved in the conduct and administration of this study as an investigator, subinvestigator, study coordinator, other study staff member, or employee of AstraZeneca, or the participant is a first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or the participant is enrolled in this study at another clinical study site.

19 Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).

20 Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

21 Previous participation in the present study.

Complete exclusion criteria are in the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2023-09-19 (Actual); Study Completion 2023-09-19 (Actual)

PRIMARY OUTCOMES:
Number and percentage of patients with adverse events | through Week 70
  Number and percentage of patients with reported adverse events.
Percentage of patients with potentially clinically significant changes in laboratory values | through Week 70
  Percentage of patients with potentially clinically significant changes in hematology, clinical chemistry, urinalysis.
Percentage of patients with potentially clinically significant changes in vital signs | through Week 70
  Percentage of patients with potentially clinically significant changes in systolic and diastolic blood pressure, temperature, respiratory rate and pulse rate.
Percentage of patients with potentially clinically significant changes in ECGs | through Week 70
  Percentage of patients with potentially clinically significant changes in 12-lead ECG recordings.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Bohannon, Study Director — AstraZeneca
Locations (14):
- United States (9):
  - Research Site, Lincoln, California
  - Research Site, Clearwater, Florida
  - Research Site, Kissimmee, Florida
  - Research Site, Lakeland, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Tampa, Florida
  - Research Site, Beachwood, Ohio
  - Research Site, Houston, Texas
- Research Site, Hamburg, Germany
- Research Site, Rzeszów, Poland
- South Africa (2):
  - Research Site, Cape Town
  - Research Site, Plumstead
- Research Site, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home